CLINICAL TRIAL: NCT02594475
Title: A Prospective, Randomized Study Comparing Efficacy and Safety Between Left Lateral Position and Prone Position for Endoscopic Retrograde Cholangiopancreatography
Brief Title: Left Lateral Position and Prone Position for Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-71
Record Dates: First submitted 2015-11-01; First posted 2015-11-03 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Choledocholithiasis
Keywords: endoscopic retrograde cholangiopancreatography, position
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Left lateral position (Experimental): Endoscopic retrograde cholangiopancreatography is performed in left lateral position in this group.
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography
- Prone position (Active Comparator): Endoscopic retrograde cholangiopancreatography is performed in prone position in this group.
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography — 1. Endoscopic retrograde cholangiopancreatography is started using conventional duodenoscope (TJF 240 or 260V, Olympus Optical Co., Ltd, Tokyo, Japan) in randomly assigned left lateral position or prone position.
  2. Selective bile duct cannulation is performed using wire-guided cannulation.
  3. In case of difficult cannulation, precut is performed using a needle-knife.
  4. After selective cannulation, cholangiogram is obtained using ERCP catheter, and endoscopic sphincterotomy and/or endoscopic papillary balloon dilation is performed.
  Other Names: Endoscopic biliary drainge

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) has been widely used in diagnosis and treatment of pancreaticobiliary diseases. Traditionally, ERCP has been performed in the prone position. The prone position for ERCP can facilitate selective bile duct cannulation, offer a better fluoroscopic image of pancreaticobiliary anatomy, and prevent aspiration of gastric contents. However, in cases of difficult in the prone position, ERCP has been performed in the left lateral or supine position. Compared with the prone position, left lateral position is more comfortable for patients, especially with limitation for cervical movement including cervical cord injury, cervical spine operation, parkinson's disease, contracture due to cerebral infarction, and allow more easy passage of the scope through the pharynx, and useful to secure airway. However, in the left lateral position, it is difficult to obtain fluoroscopic image of right hepatic duct and intrahepatic bile duct.

In cases of severe abdominal pain, severe abdominal distension, large amount of ascites, recent abdominal surgery or cervical spine surgery, intra-abdominal catheter insertion, severe obesity, it is difficult to position in prone or left lateral, therefore, ERCP may be performed in the supine position. In supine position for ERCP, there has been documented increased risk of cardiopulmonary adverse event and decreased success rate of selective bile duct cannulation.

There have been reported the efficacy and safety between the prone position and supine position for ERCP in several studies. We aimed to evaluate the efficacy and safety between the prone position and left lateral position for ERCP in this prospective, randomized study.

DETAILED DESCRIPTION:
Methods

1. Written informed consent for the endoscopic retrograde cholangiopancreatography is obtained from all patients.
2. Blood culture is performed, and intravenous 3rd generation cephalosporin is administered routinely.
3. Before endoscopic procedure, patients are randomly assigned to left lateral position or prone position for the endoscopic retrograde cholangiopancreatography.
4. Conscious sedation is performed by non-anesthesiologist-assisted method. Intravenous midazolam 0.05-0.1 mg/kg and/or intravenous propofol 0.5mg-1mg/kg is administered. Analgesics was administered intravenous meperidine 25mg in patients with older than 50 years and meperidine 50mg in patients with younger than 50 years. To limit duodenal peristalsis hyoscine-N-butylbromide is administered intravenously.
5. All patients are provided oxygen 2liter/minute via nasal prong. Patient's oxygen saturation, heart rate, blood pressure and respiration are monitored during procedure.
6. Selective bile duct cannulation is performed by wire-guided cannulation method. If adverse event is occur during endoscopic procedure, it is recorded in the case report form as intra-procedural adverse event.
7. After 4 hours, 24 hours, 2 weeks and 6 weeks of the procedure, white blood cell count, hemoglobin, platelet count, total bilirubin, aspartate transaminase, alanine transaminase, alkaline phosphatase, gamma glutamyl transaminase, amylase, lipase, abdomen X-ray, chest X-ray are performed.
8. Oral feeding is started with sips of water after 24 hours of endoscopic sphincterotomy and/or endoscopic papillary balloon dilation.
9. Development of adverse event including bleeding, perforation, pancreatitis, hyperamylasemia, infection, basket impaction, cardiopulmonary adverse event, mortality are recorded according to left lateral position or prone position for the endoscopic retrograde cholangiopancreatography.

ELIGIBILITY:
Inclusion Criteria:

* All of followings:

  1. Any of following indications for ERCP

     ① Common bile duct stone

     ② Gallstone pancreatitis

     ③ Obstructive jaundice due to malignancy (ex. Pancreas cancer, bile duct cancer, ampulla of Vater cancer)

     ④ Common bile duct invasion metastasis of other organ malignancy (ex. Hepatocellular carcinoma with bile duct invasion, metastatic lymphadenopathy with bile duct invasion from malignancy other than pancreaticobiliary malignancy)

     ⑤ Benign biliary stricture
  2. Naïve papilla
  3. Aged over 20 years

     Exclusion Criteria:
* Any of followings:

  1. History of endoscopic retrograde cholangiopancreatography
  2. Altered gastric and duodenal anatomy due to intra-abdominal surgery (ex. Billroth gastrectomy, total gastrectomy)
  3. Patients with severe infection or hemodynamic unstable (ex. septic shock, intubation, ventilator, inotropics)
  4. Recent myocardial infarction (within 6 months) or uncontrolled arrhythmia, unstable angina, or congestive heart failure
  5. Severe neurologic disease
  6. Patients with possible prone position (ex. severe abdominal pain, severe abdominal distension, large amount of ascites, recent intra-abdominal surgery, neck surgery, intra-abdominal catheter insertion, severe obesity)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2015-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
success in selective bile duct cannulation | within first 1 hour after attempt of bile duct cannulation

SECONDARY OUTCOMES:
endoscopic retrograde cholangiopancreatography-related adverse event | within 14 days after endoscopic retrograde cholangiopancreatography

CONTACTS AND LOCATIONS:
Overall Officials: Tae Young Park, Study Director — Chuncheon Sacred Heart Hospital, Hallym University College of Medicine
Locations (1):
- Hallym University Chuncheon Sacred Heart Hospital, Hallym University College of Medicine, Chuncheon, Gangwon-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ASGE Standards of Practice Committee; Maple JT, Ben-Menachem T, Anderson MA, Appalaneni V, Banerjee S, Cash BD, Fisher L, Harrison ME, Fanelli RD, Fukami N, Ikenberry SO, Jain R, Khan K, Krinsky ML, Strohmeyer L, Dominitz JA. The role of endoscopy in the evaluation of suspected choledocholithiasis. Gastrointest Endosc. 2010 Jan;71(1):1-9. doi: 10.1016/j.gie.2009.09.041. No abstract available. PMID 20105473
- [Background] Baron TH, Mallery JS, Hirota WK, Goldstein JL, Jacobson BC, Leighton JA, Waring JP, Faigel DO. The role of endoscopy in the evaluation and treatment of patients with pancreaticobiliary malignancy. Gastrointest Endosc. 2003 Nov;58(5):643-9. doi: 10.1016/s0016-5107(03)01994-1. PMID 14595292
- [Background] Costamagna G, Shah SK, Tringali A. Current management of postoperative complications and benign biliary strictures. Gastrointest Endosc Clin N Am. 2003 Oct;13(4):635-48, ix. doi: 10.1016/s1052-5157(03)00103-x. PMID 14986791
- [Background] Ferreira LE, Baron TH. Comparison of safety and efficacy of ERCP performed with the patient in supine and prone positions. Gastrointest Endosc. 2008 Jun;67(7):1037-43. doi: 10.1016/j.gie.2007.10.029. Epub 2008 Jan 18. PMID 18206877
- [Background] Froehlich F. Patient position during ERCP: prone versus supine. What about left lateral throughout? Endoscopy. 2006 Jul;38(7):755; author reply 755. doi: 10.1055/s-2006-925247. No abstract available. PMID 16810601
- [Background] Terruzzi V, Radaelli F, Meucci G, Minoli G. Is the supine position as safe and effective as the prone position for endoscopic retrograde cholangiopancreatography? A prospective randomized study. Endoscopy. 2005 Dec;37(12):1211-4. doi: 10.1055/s-2005-870511. PMID 16329019
- [Background] Tringali A, Mutignani M, Milano A, Perri V, Costamagna G. No difference between supine and prone position for ERCP in conscious sedated patients: a prospective randomized study. Endoscopy. 2008 Feb;40(2):93-7. doi: 10.1055/s-2007-995317. Epub 2007 Dec 5. PMID 18058651
- [Background] Williams EJ, Taylor S, Fairclough P, Hamlyn A, Logan RF, Martin D, Riley SA, Veitch P, Wilkinson M, Williamson PR, Lombard M; BSG Audit of ERCP. Are we meeting the standards set for endoscopy? Results of a large-scale prospective survey of endoscopic retrograde cholangio-pancreatograph practice. Gut. 2007 Jun;56(6):821-9. doi: 10.1136/gut.2006.097543. Epub 2006 Dec 4. PMID 17145737
- [Background] Owens WD, Felts JA, Spitznagel EL Jr. ASA physical status classifications: a study of consistency of ratings. Anesthesiology. 1978 Oct;49(4):239-43. doi: 10.1097/00000542-197810000-00003. PMID 697077
- [Background] Boix J, Lorenzo-Zuniga V, Ananos F, Domenech E, Morillas RM, Gassull MA. Impact of periampullary duodenal diverticula at endoscopic retrograde cholangiopancreatography: a proposed classification of periampullary duodenal diverticula. Surg Laparosc Endosc Percutan Tech. 2006 Aug;16(4):208-11. doi: 10.1097/00129689-200608000-00002. PMID 16921297
- [Background] ASGE Standards of Practice Committee; Anderson MA, Fisher L, Jain R, Evans JA, Appalaneni V, Ben-Menachem T, Cash BD, Decker GA, Early DS, Fanelli RD, Fisher DA, Fukami N, Hwang JH, Ikenberry SO, Jue TL, Khan KM, Krinsky ML, Malpas PM, Maple JT, Sharaf RN, Shergill AK, Dominitz JA. Complications of ERCP. Gastrointest Endosc. 2012 Mar;75(3):467-73. doi: 10.1016/j.gie.2011.07.010. No abstract available. PMID 22341094
- [Background] Cotton PB, Lehman G, Vennes J, Geenen JE, Russell RC, Meyers WC, Liguory C, Nickl N. Endoscopic sphincterotomy complications and their management: an attempt at consensus. Gastrointest Endosc. 1991 May-Jun;37(3):383-93. doi: 10.1016/s0016-5107(91)70740-2. PMID 2070995
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503
- [Background] Mulla SM, Scott IA, Jackevicius CA, You JJ, Guyatt GH. How to use a noninferiority trial: users' guides to the medical literature. JAMA. 2012 Dec 26;308(24):2605-11. doi: 10.1001/2012.jama.11235. PMID 23268519